CLINICAL TRIAL: NCT00248846
Title: A Randomized Trial: Changing Behavior in Post-Angioplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N01-HC-25196 (0203-694); N01HC25196 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Angioplasty Patients
Keywords: Angioplasty patients; Behavior change; Physical activity; Risk reduction
MeSH Terms: conditions — Motor Activity; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): This group received follow-up every 2-months for one year. Follow-up included questions about their heart disease progression and how well they had been able to engage in their doctor approved physical activity goal.
- Intervention Group (Experimental): This group received follow-up every 2-months for one year. Follow-up included questions about their heart disease progression and how well they had been able to engage in their doctor approved physical activity goal, which was the same as the control arm. Additionally, subjects in this arm were encouraged to use positive affect and self-affirmation techniques to motivate an increased level of participation in their physical activity goal. These subjects also received small token gifts to remind them of their study participation.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — During the physical activity goal setting process, subjects were randomly assigned to either the control or the intervention group. The intervention included receiving an additional educational workbook about using positive affect and self affirmation, as well as participating in using positive affect and self-affirmation to motivate behavior change, which in this case was to increase their physical activity level. Patient also received small token gifts to remind them of their participation in the study and to induce positive affect. The control group also set a physical activity goal and received the same follow-up, but did not participate in the positive affect and self-affirmation portion.
  Other Names: Postivie affect and self-affirmation induction vs. control
  Arms: Intervention Group

SUMMARY:
The long-term objective of this study is to determine whether a positive affect and self-affirmation condition added to an empirically demonstrated approach for motivating behavior change is more effective than a standard approach in reducing risk factor behavior among a high-risk group of patients with coronary artery disease. Thus, the goal of the project is to refine and improve strategies for long-term maintenance of physical activity among patients post-angioplasty or stent.

DETAILED DESCRIPTION:
Among coronary artery disease patients who have just had either angioplasty or stents, the objective of this randomized trial is to evaluate whether a novel behavioral intervention that employs induced positive affect and self-affirmation is more effective than an intervention without positive affect in increasing the maintenance of newly initiated physical activity post-procedure.

Secondary objectives:

* To determine whether more patients who receive the positive affect and self-affirmation intervention initiate more multiple behavior changes (e.g., changes in more health behaviors directed to their risk-factor profile) than those in the control group at one year.
* To determine whether the positive affect and self-affirmation intervention increases physical activity among patients who have depressive symptoms.
* To determine whether patients who are successful in increasing physical activity are more successful at changing other health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing coronary artery catheterization who are found to have at least single vessel stenosis and who have had revascularization with angioplasty or coronary artery stenting will be eligible for enrollment.
* Patients must be able to provide informed consent within the one week after the procedure.

Exclusion Criteria:

* Patients who are unable to walk several blocks regardless of the reason will be excluded from all the trials (e.g., arthritis, stroke, claudication).
* Enrollment in other trials designed to modify post-procedure behaviors.
* Patients who refuse to participate will be excluded.
* If at any time prior to enrollment in the study, the patient's cardiologist determines that the patient should not participate in this study, the patient will not be enrolled in the trial.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Within patient change in the Paffenbarger Exercise and Physical Activity Index | basline, at 2-month intervals(2, 4, 6, 8, 10-months) and closeout

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD

REFERENCES:
- [Background] Peterson JC, Allegrante JP, Pirraglia PA, Robbins L, Lane KP, Boschert KA, Charlson ME. Living with heart disease after angioplasty: A qualitative study of patients who have been successful or unsuccessful in multiple behavior change. Heart Lung. 2010 Mar-Apr;39(2):105-15. doi: 10.1016/j.hrtlng.2009.06.017. Epub 2009 Aug 25. PMID 20207270
- [Background] Charlson ME, Boutin-Foster C, Mancuso CA, Peterson JC, Ogedegbe G, Briggs WM, Robbins L, Isen AM, Allegrante JP; Translational Behavioral Science Research Consortium. Randomized controlled trials of positive affect and self-affirmation to facilitate healthy behaviors in patients with cardiopulmonary diseases: rationale, trial design, and methods. Contemp Clin Trials. 2007 Nov;28(6):748-62. doi: 10.1016/j.cct.2007.03.002. Epub 2007 Mar 12. PMID 17459784
- [Result] Peterson JC, Charlson ME, Hoffman Z, Wells MT, Wong SC, Hollenberg JP, Jobe JB, Boschert KA, Isen AM, Allegrante JP. A randomized controlled trial of positive-affect induction to promote physical activity after percutaneous coronary intervention. Arch Intern Med. 2012 Feb 27;172(4):329-36. doi: 10.1001/archinternmed.2011.1311. Epub 2012 Jan 23. PMID 22269589
- [Derived] Peterson JC, Charlson ME, Wells MT, Altemus M. Depression, coronary artery disease, and physical activity: how much exercise is enough? Clin Ther. 2014 Nov 1;36(11):1518-30. doi: 10.1016/j.clinthera.2014.10.003. Epub 2014 Nov 14. PMID 25456561